CLINICAL TRIAL: NCT05408208
Title: Efficacy Of Intralesional Injection Of Methotrexate Versus Triamcinolone Acetonid In Treatment Of Localized Psoriasis
Brief Title: Intralesional Injection Of Methotrexate Versus Triamcinolone Acetonid In Treatment Of Localized Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Gehad Hamdy Abdelgaber, Gehad Hamdy, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: soh-med-22-05-04
Record Dates: First submitted 2022-05-22; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Localized Psoriasis
Keywords: Intralesional Injection ,Methotrexate, localized Psoriasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Active Comparator): Intralesional injection of methotrexate
  Interventions: Drug: Intralesional Injection of Methotrexate; Drug: Triamcinolone Acetonid
- Triamcinolone Acetonid (Active Comparator): Intralesional injection of trimethinolone acetonide
  Interventions: Drug: Intralesional Injection of Methotrexate; Drug: Triamcinolone Acetonid

INTERVENTIONS:
Drug: Intralesional Injection of Methotrexate — One psoriatic lesion will treated with Intralesional injection of methotrexate (25mg /ml) at dosage of 0.1 ml /cm Another plaque will treated with intralesional ingection of distilled water as controlled plaque.
  Patients will take 6 sessions every 2 weeks for 3 months and will followed up at 2 month and 3 months after treatment .
Drug: Triamcinolone Acetonid — One lesion will treated with Intralesional injection of trimethinolone acetonide (10mg/ml) at dosage of 0.1 ml/ cm2 . another plaque will treated with Intralesional injection of distilled water as controed plaque Patients will take 6 sessions every 2 weeks for 3 months and will followed up at 2 month and 3 months after treatment .

SUMMARY:
The aim of the present study is to evaluate the efficacy of intralesional injection of methotrexate in comparison with Intralesional Injection of Triamcinolone Acetonid in localized psoriasis (body surface area < 10%) .

DETAILED DESCRIPTION:
study enrolling 30 patients of localized psoriasis. 15 patients received intralesional methotrexate :

* Taking aseptic condition ,One psoriatic plaque will treated with Intralesional injection of methotrexate (25mg /ml) at dosage of 0.1 ml /cm2.
* Another plaque will treated with intralesional ingection of distilled water as controlled plaque.
* patient will receive oral folic acid 5mg tablet every day except the day of injection.

Other 15 patients received intralesional trimethinolone acetonide:

* Taking aseptic condition , One plaque will treated with Intralesional injection of trimethinolone acetonide (10mg/ml) at dosage of 0.1 ml/ cm2 .
* another plaque will treated with Intralesional injection of distilled water as controed plaque.
* Patients will take 6 sessions every 2 weeks for 3 months and will followed up at 2 month and 3 months after treatment .

ELIGIBILITY:
Inclusion Criteria:

* patients with localized Psoriasis (body surface area<10%)

Exclusion Criteria:

* Patient refusal. Generalized psoriasis. Pregnancy. Lactation. Immunocompromised patients . Patients with history of hypersensitivity to methotrexate. Patients with other inflammatory skin disorders. Patients with chronic hepatic, renal , pulmonary ,or haematological disorders. patients on treatment for psoriasis .

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-21 (Actual); Primary Completion 2022-11-21 (Estimated); Study Completion 2023-05-21 (Estimated)

PRIMARY OUTCOMES:
Efficacy Of Intralesional Injection Of Methotrexate Versus Triamcinolone Acetonid In Treatment Of Localized Psoriasis | 3 months after treatment
  clinical and dermoscopic changes according to psoriasis area severity index

CONTACTS AND LOCATIONS:
Overall Officials: Gehad Hamdy, Principal Investigator — Gehad Hamdy Abd El-Gaber
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided